CLINICAL TRIAL: NCT01643512
Title: Heritability of Fatty Liver as Measured by MRI: a Cross Sectional Study of Twins and Family Members
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rohit Loomba, Professor, University of California, San Diego
Other Study IDs: 111282
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Liver Disease
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, plasma, urine, stool, DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most common liver disease in the United States. The cause of NAFLD is poorly defined but is thought to involve complex interactions of genetic and environmental factors. NAFLD is often associated with the traits of the metabolic syndrome including diabetes, high cholesterol or elevated blood pressure. Currently, there are no accurate noninvasive means of evaluating NAFLD and its more serious form which includes inflammation that may lead to severe scarring in the liver. The goal of this study is to evaluate shared genetic factors that underlie NAFLD and features of the metabolic syndrome as determined by blood work and radiographic studies in a cohort of twins and first degree relatives.

DETAILED DESCRIPTION:
Following an information session during which the primary consent document, a genetic sampling consent document and the UCSD HIPPA forms are reviewed, discussed and signed, the following tests and procedures will be done. For each subject, the study visit will be for 3-4 hours.

1. Subjects will undergo a detailed history, physical examination, anthropometrics and vital signs including blood pressure and pulse. Standardized questionnaires including the Alcohol Use Disorders Identification Tests (AUDIT) and Skinner Lifetime Drinking History will be used to identify alcohol use as a cause of fatty liver disease. A trained investigator will measure waist/hip ratio at the same time as other measures are taken. The Body Mass Index (BMI) will be as calculated by measuring each subject's weight (Kg) and height (m) with empty bowel and bladder and using the formula: BMI = weight (kg)/ height (m)2.
2. Blood tests: Participants will undergo phlebotomy, after an overnight fast, for complete metabolic panel (including liver function tests), complete blood count, protime, lipid panel, free fatty acids, serum insulin, hemoglobin A1C, fasting glucose, hepatitis B surface antigen, hepatitis C antibody, prothrombin time and HIV. 30ml of blood will be collected: including 5ml of serum banking, 5ml of plasma banking, 5ml of DNA banking, and 15ml for planned labs as listed above. Plasma will be stored for adipocytokines and testing of novel genes or biomarkers for NALFD in later studies. Fasting plasma glucose and plasma insulin levels will be obtained. Insulin resistance will be measured by HOMA-IR, the homeostasis assessment model of insulin resistance, where HOMA-IR (mmol/L x µU/ml) = fasting glucose (mmol/L) x fasting insulin (µU/ml)/22.5). The participants will be required to provide a stool and urine sample as well.
3. A urine pregnancy test will be performed for all women of childbearing age. Women who have had hysterectomies are excluded from pregnancy testing. If the pregnancy test is positive, the patient will not be enrolled in the study.
4. The patient will undergo magnetic resonance imaging for hepatic fat fraction.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age
2. The subject is willing and able to complete all procedures and observations specified in the protocol
3. The subject has been fully informed and has personally signed and dated the written Informed Consent/Assent and Health Insurance Portability and Accountability Act (HIPAA) provisions.

Exclusion Criteria:

1. The subject is a female who is pregnant or nursing.
2. Contraindications to MRI:

   * The subject has any contraindication to MR imaging, such as patients with pacemakers, metallic cardiac valves, magnetic material such as surgical clips, implanted electronic infusion pumps or other conditions that would preclude proximity to a strong magnetic field.
   * The subject has a history of extreme claustrophobia.
   * The subject cannot fit inside the MR scanner cavity

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twins and first degree relatives (sibling-sibling or offspring-parent).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-08; Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Loomba, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- See also: Related Info — http://gastro.ucsd.edu/fatty-liver/research/patient-research/Pages/twin.aspx